CLINICAL TRIAL: NCT01455142
Title: A Trial to Test for Bioequivalence Between NN1045 and NN5401 in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1045-3834; 2011-001569-42 (EudraCT Number); U1111-1120-3922 (Other: WHO)
Record Dates: First submitted 2011-10-17; First posted 2011-10-19 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation 1 (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- Formulation 2 (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Single injection of each formulation. The dose level will be 0.5 U/kg body weight (BW). The trial products will be administered subcutaneously (under the skin).
  Other Names: IDegAsp

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to test for bioequivalence between two formulations of insulin degludec/insulin aspart (IDegAsp) to see if the efficacy and safety obtained with formulation 1 can be assumed identical for formulation 2.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for 12 months or longer
* Body mass index from 18.0 to 28.0 kg/m^2 (both inclusive)
* HbA1c below or equal to 9.5% by central laboratory analysis

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin degludec concentration-time curve | From 0 to 120 hours after single-dose (SD)
Maximum observed serum insulin degludec concentration | After single-dose (within 0 to 120 hours after dosing)
Area under the serum insulin aspart concentration-time curve | From 0 to 12 hours after single-dose
Maximum observed serum insulin aspart concentration | After single-dose (within 0 to 12 hours after dosing)

SECONDARY OUTCOMES:
Area under the glucose infusion rate curve | From 0 to 26 hours after single-dose
Maximum glucose infusion rate | After single-dose (within 0 to 120 hours after dosing)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Graz, Austria

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com